CLINICAL TRIAL: NCT06172855
Title: The Study on the Effectiveness and Safety of Electroacupuncture at ST36 (Zusanli) in Treating Primary Premature Ejaculation
Brief Title: The Study on the Effectiveness and Safety of Electroacupuncture at ST36 in Treating Primary Premature Ejaculation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-PY-26
Record Dates: First submitted 2023-01-16; First posted 2023-12-15 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Premature Ejaculation
Keywords: Premature Ejaculation; Electroacupuncture; ST36
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Premature ejaculation (Experimental): Adult male with primary premature ejaculation. They will receive electroacupuncture at ST36 to treat premature ejaculation.
  Interventions: Device: Electroacupuncture at ST36

INTERVENTIONS:
Device: Electroacupuncture at ST36 — Electroacupuncture at ST36, which located at the anterior aspect of the lower leg, 3 cun below ST 35, one finger-breadth (middle finger) from the anterior crest of the tibia. Twice or 3 times per week, for 6 weeks.

SUMMARY:
A pilot prospective single-arm cohort study on the Effectiveness and Safety of Electroacupuncture at ST36(Zusanli) in Treating Primary Premature Ejaculation

DETAILED DESCRIPTION:
This is a pilot prospective single-arm cohort study to verify the Effectiveness and Safety of Electroacupuncture at ST36(Zusanli) in Treating Primary Premature Ejaculation, based on the result on animal study that daily electroacupuncture at ST36(Zusanli) for 30 days could delay the ejaculation of male SD rats.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60
2. Heterosexual, with a single, stable partner for more than 6 months
3. Symptoms of primary premature ejaculation: Complaints of IELT ≤ 1 min since the first sexual intercourse, and poor ability to control ejaculation leading to anxiety, annoyance, depression or/and avoidance of sexual life and other negative effects.

Exclusion Criteria:

1. Urinary system infection: Urinary tract infection symptoms (such as urinary tract irritation symptoms, prostatitis symptoms, blood semen, etc.) or urine routine shows abnormal white blood cells and red blood cells
2. Abnormal androgen: sex hormone examination shows abnormal androgen (testosterone)
3. Systemic diseases: ask about medical history of hypertension, diabetes, alcohol dependence, coronary heart disease and mental disorders
4. Organic abnormalities: Abnormal development of external genitalia, bilateral testes, epididymis and spermatic cords with obvious abnormalities on palpation
5. History of surgery and trauma: Dorsal nerve block of the penis, erectile function-related surgery, prostate surgery, pelvic surgery, etc.
6. Influence of drugs: within one month before enrollment, have taken SSRI, tramadol and other drugs to treat diseases
7. Allergy to dapoxetine and lidocaine
8. History of drug, alcohol or substance abuse in the past 6 months
9. Accompanied by erectile dysfunction: International Index of Erectile Function-5 (International Index of Erectile Function, IIEF-5) score ≤ 21 points

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline intravaginal ejaculatory latency time | Week 6, 10, 14, 18
  IELT

SECONDARY OUTCOMES:
Premature Ejaculation Diagnose Tool | Week 0, 6, 10, 14, 18
  The premature ejaculation diagnostic tool (PEDT) is a brief diagnostic measure to assess premature ejaculation
Premature Ejaculation Profile | Week 0, 6, 10, 14, 18
  Premature Ejaculation Profile (PEP) is a self-reported outcome instrument for evaluating domains of PE and its treatment and comprises of four single-item measures, a profile, and an index score.
Chinese Index of Premature Ejaculation | Week 0, 6, 10, 14, 18
  The Chinese Index of Premature Ejaculation(CIPE) has 10 questions, focusing on libido, erectile function, ejaculatory latency, sexual satisfaction and difficulty in delaying ejaculation, self-confidence and depression. Each question was responded to on a 5 point Likert-type scale.
Penile Nerve Electrophysiology | Week 0, 6, 18
  An electrophysiological technique used to examine the axonal composition and reflex activity of the penile nerve
Clinical Global Impression of Change | Week 6, 18
  Clinical Global Impressions (CGI) scale is a well-established research rating tool applicable to all psychiatric disorders that can easily be used by the practicing clinician to meet this need.
fMRI | Week 0, 6
  Measure GABA levels in thalamic regions using GABA spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Baibing Yang, Doctor, Study Chair — Nanjing Drum Tower Hospital Affiliated to Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital Affiliated to Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Serefoglu EC, McMahon CG, Waldinger MD, Althof SE, Shindel A, Adaikan G, Becher EF, Dean J, Giuliano F, Hellstrom WJ, Giraldi A, Glina S, Incrocci L, Jannini E, McCabe M, Parish S, Rowland D, Segraves RT, Sharlip I, Torres LO. An evidence-based unified definition of lifelong and acquired premature ejaculation: report of the second international society for sexual medicine ad hoc committee for the definition of premature ejaculation. Sex Med. 2014 Jun;2(2):41-59. doi: 10.1002/sm2.27. PMID 25356301
- [Background] Kimura K, Kitagawa Y, Tajima F. Effects of a Single Session of Acupuncture Treatment on Blood Pressure and Heart Rate Variability in Patients with Mild Hypertension. J Altern Complement Med. 2021 Apr;27(4):342-348. doi: 10.1089/acm.2020.0324. Epub 2021 Jan 28. PMID 33512256
- [Result] Xia JD, Chen J, Yang BB, Sun HJ, Zhu GQ, Dai YT, Yang J, Wang ZJ. Differences in sympathetic nervous system activity and NMDA receptor levels within the hypothalamic paraventricular nucleus in rats with differential ejaculatory behavior. Asian J Androl. 2018 Jul-Aug;20(4):355-359. doi: 10.4103/aja.aja_4_18. PMID 29516873
- [Result] Zhang QJ, Yang BB, Yang J, Wang YM, Dai YT, Song NH, Wang ZJ, Xia JD. Inhibitory Role of Gamma-Aminobutyric Receptors in Paraventricular Nucleus on Ejaculatory Responses in Rats. J Sex Med. 2020 Apr;17(4):614-622. doi: 10.1016/j.jsxm.2020.01.006. Epub 2020 Feb 7. PMID 32037229
- [Result] Liu S, Wang ZF, Su YS, Ray RS, Jing XH, Wang YQ, Ma Q. Somatotopic Organization and Intensity Dependence in Driving Distinct NPY-Expressing Sympathetic Pathways by Electroacupuncture. Neuron. 2020 Nov 11;108(3):436-450.e7. doi: 10.1016/j.neuron.2020.07.015. Epub 2020 Aug 12. PMID 32791039
- [Result] Sahin S, Bicer M, Yenice MG, Seker KG, Yavuzsan AH, Tugcu V. A Prospective Randomized Controlled Study to Compare Acupuncture and Dapoxetine for the Treatment of Premature Ejaculation. Urol Int. 2016;97(1):104-11. doi: 10.1159/000445253. Epub 2016 Apr 7. PMID 27049323
- [Result] Lu MJ, Yu Z, He Y, Yin Y, Xu B. Electroacupuncture at ST36 modulates gastric motility via vagovagal and sympathetic reflexes in rats. World J Gastroenterol. 2019 May 21;25(19):2315-2326. doi: 10.3748/wjg.v25.i19.2315. PMID 31148903